CLINICAL TRIAL: NCT01739244
Title: Dose Finding Clinical Trial With SYL040012 to Evaluate the Tolerability and Effect on Intraocular Pressure in Subjects With Ocular Hypertension or Open Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sylentis, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYL040012_III
Record Dates: First submitted 2012-11-12; First posted 2012-12-03 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
Keywords: Glaucoma; Open Angle Glaucoma; Ocular Hypertension; IOP; RNAi; siRNA; beta inhibitor
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SYL040012 eye drops dose A (Experimental): Ocular topical administration of SYL040012 eye drops dose A
  Interventions: Drug: SYL040012
- SYL040012 eye drops dose B (Experimental): Ocular topical administration of SYL040012 eye drops dose B
  Interventions: Drug: SYL040012
- SYL040012 eye drops dose C (Experimental): Ocular topical administration of SYL040012 eye drops dose C
  Interventions: Drug: SYL040012
- Placebo (Placebo Comparator): Ocular topical administration of placebo eye drops
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYL040012 — Ocular topical administration of SYL040012 for 14 consecutive days
  Arms: SYL040012 eye drops dose A; SYL040012 eye drops dose B; SYL040012 eye drops dose C
Drug: Placebo — Ocular topical administration of placebo for 14 consecutive days
  Arms: Placebo

SUMMARY:
The aim of this dose-finding clinical trial is to evaluate the systemic tolerability, local tolerability and intraocular pressure lowering effect of three different doses of SYL040012 in subjects with ocular hypertension or open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide signed informed consent prior to participation in any study-related procedures.
* Male and female subjects in good or fair general health as assessed by the investigator.
* ≥18 years of age.
* Previous history or newly diagnosed elevated IOP (≥21 mmHg) with or without open-angle glaucoma in both eyes.
* Normal result, or result typical for open-angle glaucoma of the following assessments in both eyes or available results in writing within the last 3 months prior to baseline period i.e. up to 4 months before Day 1, on condition that no new ocular signs or symptoms (e.g. marked deterioration of vision, eye pain) has occurred since then which would justify a repeat examination:
* Visual field 24-2 or equivalent
* Optical coherence tomography (OCT)
* Best corrected visual acuity ≥0.5 (20/40) on the Snellen chart, or ≤ 0.3 logMAR
* Schirmer test (lacrimation)
* Funduscopy

Exclusion Criteria:

* Pregnant or breastfeeding females or those with a positive pregnancy test. Females of childbearing potential who will not use a medically acceptable contraceptive method from selection and during the hole study.
* Females of childbearing potential not willing to use a medically acceptable contraceptive method from enrolment until after the follow-up visit.
* Any current disease or condition that might compromise the respiratory, cardiovascular, endocrine, neurological, haematological, renal, or gastrointestinal function.
* Previous chronic processes or with rebound characteristics that could interfere with the study according to the investigator's judgment.
* Body temperature.
* Intolerability of any components of SYL040012 or placebo.
* Unable to comply with the clinical trial requirements as judged by the investigator.
* Beta blockers or corticosteroids use (other than cutaneous or intra-articular) for the treatment of concurrent diseases, even if sporadically, or any ocular or nasal vasoconstrictor treatment in the last 15 days prior to the first investigational product administration
* Previous refractive surgery; cataract extraction in the last 6 months
* Previous surgery for glaucoma.
* Participation in a clinical trial within 2 months before the enrolment visit
* Use of any other investigational product within 60 days before the enrolment visit.
* Other drugs for the treatment of concurrent diseases are allowed. However, their dosages should be kept constant throughout the study.
* Use of contact lenses in the last 7 days prior to the first investigational product administration and wearing contact lenses throughout the trial
* History of ocular infection or inflammation within the last 3 months before the enrolment visit
* Angle-closure or pigmentary glaucoma.
* Chronic or current acute eye diseases such as scleritis, uveitis, blepharitis, conjunctivitis, or ocular Herpes simplex virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Difference in AUC between IOP Curve Obtained at the Established Time Points and the Same Curve Performed at Baseline Period | 14 days + (4-7 days)
Simple Corneal and Conjunctival Evaluation | 15 days + (3-6 days)

SECONDARY OUTCOMES:
Visual acuity, anterior segment and ocular fundus examination as measures of local tolerability. | 14 days + (4-7 days)
Physical exploration and laboratory tests as measurements of general tolerability | 14 days + (4-7 days)
Assessment of Adverse Events Appearance | 14 days + (4-7 days)

CONTACTS AND LOCATIONS:
Locations (11):
- Estonia (2):
  - East Tallin Central Hospital, Tallinn
  - Eye Clinic Dr. Krista Turman, Tallinn
- Germany (3):
  - Uniklinik Köln, Cologne
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Mainz, Mainz
- Spain (6):
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Institut Català de Retina, Barcelona
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Instituto de Oftalmobiología Aplicada, Valladolid